CLINICAL TRIAL: NCT04510740
Title: JADE - Clinical Research Platform on Treatment and Outcome in Patients With Hepatocellular or Cholangiocellular Cancer
Brief Title: Liver Cancer Registry Platform
Acronym: JADE
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-100425
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma (HCC); Cholangiocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hepatocellular Carcinoma (HCC): Patients with Hepatocellular Carcinoma (HCC)
  Interventions: Other: Physician's choice according to patient's needs.
- Cholangiocarcinoma (CCC): Patients with Cholangiocarcinoma (CCC)
  Interventions: Other: Physician's choice according to patient's needs.

INTERVENTIONS:
Other: Physician's choice according to patient's needs. — Routine care as per site standard.

SUMMARY:
The purpose of the project is to set up a national, prospective, longitudinal, multicenter cohort study with associated satellites, a tumor registry platform, to document uniform data on characteristics, molecular diagnostics, treatment and course of disease, to collect patient-reported outcomes and to establish a decentralized biobank for patients with Hepatocellular Carcinoma (HCC) or Cholangiocarcinoma (CCC) in Germany.

DETAILED DESCRIPTION:
JADE is a national, observational, prospective, longitudinal, multicenter cohort study (tumor registry platform) with the purpose to record information on the antineoplastic treatment of HCC or CCC in Germany. The registry will follow patients for up to three years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

Health-related quality of life in patients with HCC / CCC will be evaluated for up to three years.

ELIGIBILITY:
Inclusion criteria:

* Confirmed hepatocellular carcinoma (HCC) or cholangiocarcinoma (CCC) als early, intermediate or advanced/metastatic stage
* Age ≥ 18 years
* Signed and dated informed consent (IC):

  * For participation in the PRO module: Before primary locoregional therapy or start of first systemic treatment
  * For no participation in the PRO module: No later than 8 weeks after primary locoregional therapy or start of first systemic treatment

Exclusion criteria:

Patients treated with best supportive care (BSC) only (i.e. no surgery, no radiotherapy, no ablative procedures, no systemic anti-tumoral therapies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with hepatocellular carcinoma (HCC), or cholangiocarcinoma (CCC) starting treatment for early, intermediate or advanced disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Course of treatment (treatment reality). | 3 years per patient.
  Documentation of anamnestic data and therapy sequences.

SECONDARY OUTCOMES:
Best Response. | 3 years per patient.
  Documentation of response rates per line of treatment.
Progression-free survival. | 3 years per patient.
  Documentation of progression-free survival per line of treatment.
Overall survival. | 3 years per patient.
  Documentation of overall survival per line of treatment.
Health-related quality of life (Patient-reported outcome, PRO). | 3 years per patient.
  EORTC QLQ-C30 core questionnaire [European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire; Scale 0-100; a high scale score represents a higher response level: (a) global health status: a high score represents high quality of life, (b) functional scales: a high score represents high/healthy level of functioning, (c) symptom scales/items: a high score represents high level of symptomatology or problems]
Carcinoma Health-related quality of life (Patient-reported outcome, PRO). | 3 years per patient.
  EORTC QLQ-HCC18, the hepatocellular carcinoma specific module / EORTC QLQ-BIL21, the cholangiocarcinoma specific module [European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire; Scale 0-100; a high score for scales and single items represents a high level of symptomatology or problems].

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berg, Prof.Dr., Study Chair — Leipzig; Peter R. Galle, Prof.Dr., Study Chair — Mainz; Wolf P. Hofmann, Prof.Dr., Study Chair — Berlin; Achim Kautz, Study Chair — Köln; Philippe Pereira, Prof.Dr., Study Chair — Heilbronn; Karin Potthoff, Dr., Study Chair — Freiburg im Breisgau; Jan Schröder, PD Dr., Study Chair — Mülheim an der Ruhr; Robert Thimme, Prof.Dr., Study Chair — Freiburg im Breisgau
Locations (1):
- Multiple sites all over germany, Multiple Locations, Germany